CLINICAL TRIAL: NCT06315257
Title: A Randomized, Open-label Clinical Trial to Assess the Safety, Feasibility and Immunogenicity of Adjuvant PVX7 Immunotherapy Regimens in Advanced Cervical Cancer Patients
Brief Title: A Clinical Trial to Assess PVX7 Immunotherapy Regimens in Advanced Cervical Cancer Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J23105sIRB; IRB00388854 (Other: Johns Hopkins)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, TA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pBI-11 DNA plus TA-HPV via Skin Scarification (Experimental): Participants will receive pBI-11 DNA and TA-HPV via Skin Scarification
  Interventions: Drug: PVX7
- pBI-11 DNA plus TA-HPV via IM Injection (Experimental): Participants will receive pBI-11 DNA and TA-HPV via IM Injection
  Interventions: Drug: PVX7

INTERVENTIONS:
Drug: PVX7 — PVX7 Immunotherapy
  Other Names: pBI-11 DNA + TA-HPV

SUMMARY:
A Feasibility Trial of PVX7 vaccine in advanced cervical cancer patients who have completed primary definitive therapy.

DETAILED DESCRIPTION:
A Feasibility Trial of PVX7 in advanced cervical cancer patients who have completed primary definitive therapy.

* Safety and immunogenicity study
* Patients are randomized in a 1:1 ratio to two cohorts, up to 16 patients in each of intramuscular or skin scarification vaccine injection, up to 32 patients total
* Human Immunodeficiency Virus (HIV)-negative patients only
* Treatment dose: Arm A: pBI-11 DNA (3 mg) twice via intramuscular (IM) injection, followed by one dose of TA-HPV (2.5x105 pfu) via skin scarification; Arm B: pBI-11 DNA (3 mg) twice, followed by one dose of TA-HPV (107 pfu) via IM injection
* Schedule for administration: PVX7 vaccination at weeks 1, 5, and 9
* Follow-up for 2 years per standard of care (SoC)

ELIGIBILITY:
Inclusion Criteria:

* Female subjects age 18 years or older with diagnosis of advanced (stage IB1-IVA) cervical cancer and have completed primary treatment (consisting of any of the following as per NCCN guideline standard of care: surgical resection, radiation, and/or platinum-based chemotherapy) within the past 12 months.

Patients who are recommended to receive anto-PD-1 or anti-PD-L1 therapy after chemoradiation are eligible to enroll and can continue to receive such therapy while receiving study drug.

* No history of or current evidence of residual disease or disease recurrence based on imaging and clinical assessments within 8 weeks of enrollment
* HIV uninfected
* Hepatitis B surface antigen negative
* Anti-hepatitis C (HCV) antibody negative or negative HCV polymerase chain reaction (PCR)
* Patients who are able and willing to comply with all study procedures and voluntarily sign an informed consent form
* Adequate organ function as defined by the following parameters:
* white blood cell count ≥ 3,000
* lymphocyte number ≥ 500
* absolute neutrophil count ≥ 1,000
* platelets ≥ 90,000
* hemoglobin ≥ 9
* total bilirubin <1.5 X upper limit of normal (ULN), <3 x ULN if Gilbert's disease
* Aspartate Transferase(AST)/Alanine Transaminase (ALT) <3 X ULN
* creatinine < 1.5 X ULN or estimated creatinine clearance ≥ 60 ml/min per Modified Cockcroft-Gault Formula
* Eastern Cooperative Oncology Group performance status of 0 or 1
* All clinically significant toxicities related to prior therapy should be less than or equal to Grade 1 at time of enrollment
* Ability and willingness for one month post vaccination to follow vaccine inoculation site care and avoid close social contact with children under 1 year old or close social or domestic contact with a pregnant woman or individuals at high risk of serious adverse effects of vaccinia virus, for instance, those with past or present eczema, or immunodeficiency states including HIV infection

Exclusion Criteria:

* Women of child-bearing potential (i.e., those who have had fertility-sparing procedures for the management of cervical cancer) will be excluded unless agreed to remain sexually abstinent or have a partner who is sterile (i.e. vasectomy), or use methods of contraception (e.g., oral contraception, barrier methods, spermicide, intrauterine device (IUD)), throughout the first 6 months of the study.
* Because there is a risk for adverse events in nursing infants, breastfeeding must be discontinued if the mother is treated on study.
* Diagnosed with a recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; patients diagnosed with acquired, hereditary, or congenital immunodeficiencies
* Diagnosis with a medical condition that requires systemic treatment with immunosuppressive drugs such as cyclosporine, adrenocorticotropic hormone (ACTH), alkylating agents, antimetabolites, radiation, Tumor Necrosis Factor (TNF) inhibitors, or systemic corticosteroids, either chronically or within 30 days of first PVX7 vaccination.
* Administration of any blood product within 30 days of signing informed consent.
* Need for ongoing therapeutic anticoagulation during the study period due to concern for increased risk of bleeding.
* Previous severe allergic reaction or hypersensitivity to a vaccine or any of its components
* Participation in a study with an investigational compound or device within 30 days of signing informed consent
* History of seizures (unless seizure free for 5 years)
* Known active central nervous system disease
* Surgery within 30 days of first PVX7 vaccination, excluding minor procedures
* Diagnosis with an uncontrolled intercurrent illness including, but not limited to, ongoing, or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Diagnosis with an active autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), ankylosing spondylitis)
* History of myocarditis or pericarditis.
* Known underlying heart disease (e.g., cardiomyopathy, congestive heart failure, symptomatic arrhythmia not controlled by medication, unstable angina, history of acute myocardial infarction or cerebrovascular accident within the past 6 months).
* Patients and the patients close social, sexual, or domestic contacts may not have non-healed wounds or active exfoliative skin conditions such as: Eczema, Burns, Impetigo, Varicella-zoster virus infection, Herpes simplex virus infection, Severe acne, Severe diaper dermatitis with extensive areas of denuded skin, Psoriasis, Lichen planus, Darier disease (keratosis follicularis).
* History or presence of atopic dermatitis
* Inability or unwillingness to for one month post vaccination follow vaccine inoculation site care and avoid social contact with children under 1 year old or close social or domestic contact with a pregnant woman or individuals at high risk of serious adverse effects of vaccinia virus, for instance, those with past or present eczema, or immunodeficiency states including HIV infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals with a cervix
Enrollment: 32 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Safety of PVX7 as assessed by adverse events | 12 months
  To assess the safety of PVX7 immunotherapy to patients with advanced cervical cancer who have completed primary therapy by evaluating Adverse Events (AEs).
Feasibility of PVX7 | 12 months
  To assess the feasibility of PVX7 immunotherapy to patients with advanced cervical cancer who have completed primary therapy. Feasibility is measured by the ability of patients to receive all three doses of vaccine.

SECONDARY OUTCOMES:
Cellular Immune Response | 12 months
  To evaluate the systemic Human Papillomavirus (HPV)16/18 E6/E7-specific cellular immune responses to PVX7 immunotherapy by measuring the number of interferon gamma+ Cluster of Differentiation (CD)8 Tcells/mL with overlapping peptides covering HPV16/18 E6/E7 protein
Immune Response | 12 months
  To compare the route of administration associated with the greatest immune response in patients with advanced cervical cancer who have completed primary standard of care treatment
Presence of circulating HPV DNA | 12 months
  Measure presence of circulating HPV DNA load in blood pre- and post-PVX7 immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gaillard, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared with NIH and other participating site.